CLINICAL TRIAL: NCT05535699
Title: Scapular Muscle Strengthening Versus Scapular Proprioceptive Neuromuscular Facilitation In Shoulder Impingement Syndrome
Brief Title: Scapular ms Strength vs PNF in SIS Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: finishing some devices
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, amr mohamed ahmed khalil, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS strength VS PNF IN SIS
Record Dates: First submitted 2022-08-29; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Impingement
Keywords: pnf
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- scapular muscle strengthening exercises (Experimental): Group A (n=22): will receive a program of scapular muscle strengthening exercises for 18 sessions (3 sessions per week for six weeks)
  Interventions: Other: exercises
- PNF exercise (Experimental): Group B (n=22): will receive a scapular PNF exercise program for the same frequency as in group A
  Interventions: Other: exercises
- control (No Intervention): Group C (n=22): will be a control group who will not receive any treatment during the study period.

INTERVENTIONS:
Other: exercises — scapular exercise
  Arms: PNF exercise; scapular muscle strengthening exercises

SUMMARY:
HYPOTHESES:

1. There will be no significant difference between scapular muscle strengthening and PNF exercise on improving muscle strength of upper trapezius in patients with shoulder impingement syndrome.
2. There will be no significant difference between scapular muscle strengthening and PNF exercise on improving muscle strength of middle trapezius in patients with shoulder impingement syndrome.
3. There will be no significant difference between scapular muscle strengthening and PNF exercise on improving muscle strength of lower trapezius in patients with shoulder impingement syndrome.
4. There will be no significant difference between scapular muscle strengthening and PNF exercise on improving muscle strength of serratus anterior in patients with shoulder impingement syndrome.
5. There will be no significant difference between scapular muscle strengthening and PNF exercise on muscle ratio of upper trapezius/lower trapezius muscles in patients with shoulder impingement syndrome.
6. There will be no significant difference between scapular muscle strengthening and PNF exercise on muscle ratio of upper trapezius/middle trapezius muscles in patients with shoulder impingement syndrome.
7. There will be no significant difference between scapular muscle strengthening and PNF exercise on muscle ratio of upper trapezius/serratus anterior muscles in patients with shoulder impingement syndrome.
8. There will be no significant difference between scapular muscle strengthening and PNF exercise on scapular symmetry at 0⁰ abduction in patients with shoulder impingement syndrome.
9. There will be no significant difference between scapular muscle strengthening and motor control exercise on scapular symmetry at 45⁰ abduction in patients with shoulder impingement syndrome.
10. There will be no significant difference between Scapular muscle strengthening and motor control exercise on scapular symmetry at 90⁰ abduction in patients with shoulder impingement syndrome.
11. There will be no significant difference between scapular muscle strengthening and PNF exercise on improving pain in patients with shoulder impingement syndrome.
12. There will be no significant difference between scapular muscle strengthening and PNF exercise on improving function in patients with shoulder impingement syndrome.

DETAILED DESCRIPTION:
Sub-acromial Impingement Syndrome (SIS) has been identified with a prevalence of almost 40% among shoulder pathologies. SIS has significant economic consequences owing to its treatment costs and losses incurred through workplace absenteeism.

Alterations in scapular muscle performance have been found in subjects with scapular dyskinesis. Hyperactivity of the upper trapezius (UT) with reduced middle (MT) and lower trapezius (LT) muscle activation in addition to insufficient serratus anterior (SA) muscle function have been related to decreased amounts of scapular upward rotation, external rotation, and posterior tilt in patients .

Research into scapular stability exercises for the management of SIS is increasing, yet there is little evidence on their efficacy .

The addition of scapular stabilization exercises to stretching and strengthening exercises can be significantly beneficial in increasing the strength, developing joint position sense and decreasing dyskinesia.

Proprioceptive neuromuscular facilitation (PNF) is a rehabilitation concept which is widely used by physical therapists , promoting motor learning, motor control, strength and mobility . This comprehensive rehabilitation approach includes task-oriented training with manual facilitation aimed at motor learning and motor control .

To the authors' knowledge, none of the studies has investigated the potential effect abnormal scapular muscle strengthening versus PNF exercise on the muscle strenth, muscle ratio, and ROM of the scapula during arm elevation in patient with SIS.

ELIGIBILITY:
Inclusion Criteria:

* • age of 20-50 years.

  * body mass index (BMI)<20 kg/m2
  * subjects complaining Shoulder impingement.
  * subjects with altered scapular resting positions and dyskinesis (
  * Subjects will be included if they met at least 2 of the following 5 criteria: Neer's Impingement Test, Hawkins-Kennedy Impingement Test, Supraspinatus ("Empty Can" or Jobe) Test, Apprehension and relocation Tests

Exclusion Criteria:

* Undergone shoulder surgery.
* exhibited symptoms related to the cervical spine.
* taking nonsteroidal anti-inflammatory medications.
* received a steroid injection in the past 12 months.
* were already enrolled in a physical therapy program.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-09-12 (Estimated); Primary Completion 2023-04-12 (Estimated); Study Completion 2023-04-12 (Estimated)

PRIMARY OUTCOMES:
muscle strength for scapular muscles by Lafayette hand held dynamometer | baseline
  muscle strength of upper trapezius,middle trapezius ,lower trapezius and serratus anterior in patients with shoulder impingement syndrome. pre and post application of between scapular muscle strengthening and PNF exercise
muscle ratio by dividing muscle strength of each muscle on the other | baseline
  muscle ratio of upper trapezius/lower trapezius,upper trapezius/middle trapezius and upper trapezius/serratus anterior muscles in patients with shoulder impingement syndrome. pre and post application of between scapular muscle strengthening and PNF exercise
muscle angle by lateral scapular slide test | baseline
  scapular symmetry at 0⁰ abduction ,45⁰ abduction and 90⁰ abduction in patients with shoulder impingement syndrome pre and post application of between scapular muscle strengthening and PNF exercise

SECONDARY OUTCOMES:
pain improvement by shoulder pain and disability index. | baseline
  improving pain in patients with shoulder impingement syndrome.
function improvment by shoulder pain and disability index. | baseline
  improving function in patients with shoulder impingement syndrome pre and post application of between scapular muscle strengthening and PNF exercise

CONTACTS AND LOCATIONS:
Overall Officials: mohamed AH ABDELMEGEED, lecturer, Study Director — Cairo University; salwa fadl, PROFESSOR, Study Chair — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aceituno-Gomez J, Garcia-Madero VM, Blazquez-Gamallo R, Harto-Martinez AM, Mohedano A, Vinuela A, Avendano-Coy J, Gomez-Soriano J, Munoz-Gonzalez A, Gonzalez-Gonzalez J, Criado-Alvarez JJ. [Health-related quality of life in patients diagnosed with subacromial syndrome in the Talavera Integrated Area]. Rev Esp Salud Publica. 2019 Oct 17;93:e201910094. Spanish. PMID 31621693

DOCUMENTS (1):
  • Study Protocol (2022-05-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT05535699/Prot_000.pdf